CLINICAL TRIAL: NCT04731818
Title: An Exploratory Phase 1 Mechanism-of-action Study of ZB-06, a Vaginal Film Containing HC4-N, an Anti-sperm Monoclonal Antibody.
Brief Title: An Exploratory Study of ZB-06 as a Vaginal Contraceptive Film
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: KBio Inc (Industry)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZB-06-01
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: This is a Phase 1a, single center, open-label, crossover, mechanism of action and proof of concept study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZB-06 (Experimental): All participants will receive a single ZB-06 film for intravaginal administration prior to intercourse.
  Interventions: Biological: ZB-06

INTERVENTIONS:
Biological: ZB-06 — ZB-06 is a polyvinyl alcohol-based film containing 20 mg of human contraceptive antibody (HCA) for topical intravaginal administration.

SUMMARY:
This is an early Phase 1 study to establish proof-of-concept by determining whether an intravaginal film containing a human contraceptive antibody (ZB-06) shows promise to provide contraceptive efficacy using the post-coital test, a surrogate measure of efficacy. The study will also evaluate the safety and pharmacokinetics of ZB-06.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 50 years, inclusive
* General good health, by volunteer history and per investigator judgment
* History of regular menstrual cycles of 21 - 35 days (inclusive), by volunteer report
* History of a normal PAP smear or ASCUS with negative HPV testing within the previous 12 months
* Willing to abstain from intercourse and use of vaginal medications, lubricants, and other products as required in the protocol
* Willing to use non-spermicidal, lubricated condoms for any vaginal intercourse from the first day of each menstrual cycle until 72 hours before expected midcycle
* In a mutually monogamous relationship with a male partner who:

  * Is at least 18 years old
  * Has no known risk for sexually transmitted infections (STIs)
  * Is willing and able to comply with protocol requirements including sexual activity/ abstinence and condom use requirements
  * Can engage in vaginal intercourse with the participant, with and without condoms, as specified in protocol
* Protected from pregnancy by female surgical sterilization
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy genital tract sample collection
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* History of hysterectomy
* Surgical sterility or known history of infertility in male partner
* Sterility or known history of sperm dysfunction in male partner
* Currently pregnant by urine pregnancy test at the enrollment visit, or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome
* Current use of any hormonal contraceptive or a copper or hormonal IUD, or use of Depo-Provera in the last 120 days
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* Significant gynecological abnormalities (including abnormal vaginal bleeding, excessive vaginal discharge, or vulvar/vaginal pain or irritation)
* Current UTI, vaginal candidiasis, or symptomatic bacterial vaginosis
* History of sensitivity/allergy to ZB-06 film components, for either the volunteer or her male partner
* In the last three months, either the volunteer or her male partner diagnosed with or treated for any STI or pelvic inflammatory disease, or either partner with known risk factors for sexually transmitted infections. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, or HIV at the screening visit
* Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for an STI
* Known current drug or alcohol abuse which could impact study compliance
* Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or her male partner which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will enroll 15 couples comprised of women in monogamous heterosexual relationships with male partners.
Enrollment: 20 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

REFERENCES:
- [Derived] Thurman AR, Moench TR, Hoke M, Politch JA, Cabral H, Mausser E, Nador E, Morton J, Hamorsky K, Swope K, Bratcher B, Anderson DJ, Whaley KJ. ZB-06, a vaginal film containing an engineered human contraceptive antibody (HC4-N), demonstrates safety and efficacy in a phase 1 postcoital test and safety study. Am J Obstet Gynecol. 2023 Jun;228(6):716.e1-716.e12. doi: 10.1016/j.ajog.2023.02.024. Epub 2023 Mar 2. PMID 36870409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ZB-06
Started | 20
Completed | 8
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Data from participants who completed both the baseline and the product PCT study visits
Arm/Group | ZB-06
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (5.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants that completed baseline and product PCT visits
  Participants
    Hispanic or Latino | 2
    Not Hispanic or Latino | 6
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants that completed baseline and product PCT visits
  Participants
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 5
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Surrogate Contraceptive Efficacy
Description: Number of progressively motile sperm in aspirated endocervical mucus when using ZB-06 prior to intercourse.
Time Frame: 2-3 hours after sexual intercourse.
Population: Data from all participants who complete both the baseline and the product use post coital test visits
Measure: Mean (Standard Deviation); unit: sperm per high power field
Arm/Group | ZB-06
Number analyzed (Participants) | 8
sperm per high power field
  Baseline Post Coital Test | 25.86 (30.58)
  Product Use Post Coital Test | 0.04 (0.06)
  Post Product Use Post Coital Test | 47.39 (37.43)
Statistical Analysis 1: Comparison: ZB-06; Test type: Superiority; p < 0.0001, ANOVA — analyzed by 1-way repeated measures analysis of variance (ANOVA) with post hoc Tukey multiple comparison test; 1 way repeated measures ANOVA; Mean Difference (Final Values) = 0.0001

2. Secondary Outcome: Adverse Events
Description: Incidence of Grade 2 or Greater Adverse Events during product use versus during baseline observation.
Time Frame: Baseline through study exit encompassing a minimum of three menstrual cycles of 21-35 days.
Population: Assess the incidence of Grade 2 or greater adverse events (AEs) in the participant and/or her male partner in the interval between baseline visit 4 and visit 6.
Measure: Count of Units; unit: Number of TEAEs
Units Other Than Participants: Number of TEAEs
Arm/Group | ZB-06
Number analyzed (Participants) | 8
Number analyzed (Number of TEAEs) | 1
Number of TEAEs
  Product use | 1
  Post Product Use | 0

ADVERSE EVENTS:
Time Frame: AE event monitoring for this study will began at the time of informed consent (Visit 1) through the last (visit 10), on average 3 months. First Screening was conducted February 8, 2021, and last subject last visit was February, 24, 2022.
Description: From the time of informed consent to last visit
Arm/Group | ZB-06
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZB-06 (N=8)
Hyperkalemia (Renal and urinary disorders) | 1 (1) — One TEAE, a critically high serum potassium level (6.8 mEq/L), was detected during the screening visit test was repeated and the serum potassium value was normal at 5.2 mEq/L. Deemed not related to study product or procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04731818/Prot_SAP_000.pdf